CLINICAL TRIAL: NCT06456996
Title: Population Medicine Multimorbidity Interventions in Xishui on a High-Risk COPD Population: a Cluster Randomized Controlled Trial
Brief Title: Impact of Multi-Component Interventions on High Risk COPD Population
Acronym: POPMIX-COPD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College (Other)
Collaborators: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Simiao Chen, Professor, Peking Union Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CAMS&PUMC-IEC-2024-040
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-06

CONDITIONS: Multimorbidity; Population Medicine; Chronic Obstructive Pulmonary Disease
Keywords: Multi-component intervention for multimorbidity; Population Medicine; Clustered RCT; High-risk COPD population
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): Within the intervention arm, all medical practitioners will be under a pay-for-population mechanism to incentivize them to care for the overall population health within their township. For High-risk COPD population in the intervention arm, we provide community-based spirometry pulmonary function test (PFT) and education; If individuals whose post-bronchodilator FEV1/FVC<0.7, they will be spirometry-defined COPD patients and will be encouraged to seek treatment and medication to the superior hospitals. Additionally, we provide (1) two digital health intervention programs to smokers and individuals with mental health issues; (2) CBT-based health education for study participants with abnormal BMI; (3) active recruitment into National Essential Public Health Program in China for those with abnormal blood pressure and blood glucose. Intensive follow-ups will be conducted at month 3 (telephone interview), month 6 (face-to-face with full steps of physical examination), and month 12.
  Interventions: Combination Product: Multi-component intervention package
- Control Arm (No Intervention): Those who are assigned in the control arm, we will ask them to finish the same COPD-SQ online questionnaire with notification of his or her COPD high risk status and a face-to-face survey. No physical examinations, community-based pulmonary function tests will be given at baseline. However, at month 12, we will provide community-based pulmonary function tests and physical examinations besides face-to-face survey.

INTERVENTIONS:
Combination Product: Multi-component intervention package — 1. Community-based spirometry pulmonary function tests and result interpretations and health education for COPD;
  2. A digital health intervention program, NicQuit, for smokers(very familiar with intelligent mobile phone);
  3. A digital health intervention program, EmoEase, for individuals whose WEMWBS questionnaire score is lower than 45(very familiar with intelligent mobile phone);
  4. Health education to smokers for smoking cessation;
  5. Health education to individuals with mental health issues;
  6. Encouragement to seek professional medication treatment in superior hospitals for spirometry-defined COPD patients;
  7. To actively include individuals whose blood pressurei s higher than 140/90 mmHg or/and whose random blood glucose higher than 11.1 mmol/L into the National Essential Public Health Service in China;
  8. A CBT-based health education to the BMI abnormal, i.e., BMI > 24.0 or BMI < 18.5;
  9. Pay-for-population mechanism for medical practitioners.
  Arms: Intervention arm

SUMMARY:
Study Participants: High-risk COPD population, defined as individuals whose score of COPD-SQ is 16 and above and whose age is 35 and above. COPD-SQ questionnaire will be assigned to a representative sample of local residents in Xishui County, and they will finish the questionnaire online through mobile phone.

Intervention: Within the intervention arm, we have constructed a population-based pay-for-performance mechanism to encourage medical practitioners to care for population health. For study participants in the intervention arm, we will ask them to finish an online COPD-SQ questionnaire with notification of his or her COPD high risk status. Those whose score exceeds 16 will be invited to do a face-to-face survey, simple physical examination, pulmonary function tests, and provide a multi-component intervention at baseline. For High-risk COPD population in the intervention arm, we provide community-based spirometry pulmonary function test (PFT) and education; If individuals whose post-bronchodilator FEV1/FVC<0.7, they will be spirometry-defined COPD patients and will be encouraged to seek treatment and medication to the superior hospitals. Additionally, we provide (1) two digital health intervention programs to smokers and individuals with mental health issues; (2) CBT-based health education for study participants with abnormal BMI; (3) active recruitment into National Essential Public Health Program in China for those with abnormal blood pressure and blood glucose. Intensive follow-ups will be conducted at month 3 (telephone interview), month 6 (face-to-face with full steps of physical examination), and month 12.

Comparison: Those who are assigned in the control arm, we will ask them to finish the same COPD-SQ online questionnaire with notification of his or her COPD high risk status and a face-to-face survey. No physical examinations, community-based pulmonary function tests will be given.

Outcomes: The primary outcomes are COPD knowledge, COPD screening, and FEV1 measurement at month 12.

ELIGIBILITY:
Inclusion Criteria:

* Aged 35 and above;
* COPD-SQ score is 16 and above;
* Residents who have lived in one township over the past 3 months and plan to reside in the same township in the upcoming year;
* Finished the informed consent.

Exclusion Criteria:

* Pregnancy and other conditions that are not allowed to finish pulmonary function tests;
* Severe cognitive disorder or total loss of capability of daily living

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7400 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Chronic Diseases Controlled | 1 year
  Among all objectively measured health conditions and diseases (COPD, asthma, BMI, hypertension, Type 2 diabetes, depression symptoms, anxiety symptoms), the number of chronic diseases controlled defined by objective measurement at month 12.
Lung function testing | 1 year
  Definition: Have you ever had a pulmonary function test?; Variable type: Binary; Measurement: Respondent's answer to the question;
FEV1 measurement | 1 year
  Definition: Forced Expiratory Volume in one second (FEV1); Variable type: Continuous; Measurement: Pulmonary function test, portable spirometry;

SECONDARY OUTCOMES:
Self-rated health status | 1 year
  Definition: General self-assessed health status; Variable type: Continuous; Measurement: EQ-5D-5L scale; Introduction to EQ-5D-5L scale: The 5-level EQ-5D version (EQ-5D-5L) was introduced by the EuroQol Group in 2009 to improve the instrument's sensitivity and to reduce ceiling effects, as compared to the EQ-5D-3L. The scale could be transferred to health utility value, ranging from 0 to 1 continuously. 0 represents death and 1 represents perfect health
COPD knowledge | 1 year
  Definition: Excerpt from COPD-KQ, selecting questions that test the COPD knowledge for population; Variable type: Continuous; Measurement: COPD-KQ excerpt; Introduction to COPD-KQ excerpt: An excerpt from COPD knowledge questionnaire, which contains 9 questions which we consider could be beneficial to general population to enhance the common knowledge of COPD. Minimum value is 0 and maximum value is 9, the higher the value, the more correct statements one has chosen.
Self-awareness of COPD | 1 year
  Definition: Have you ever been diagnosed with COPD?; Variable type: Binary; Measurement: Respondent's answer to the question;
COPD treatment adherence | 1 year
  Definition: Are you currently receiving a COPD treatment plan prescribed by a doctor or other healthcare professional?; Variable type: Binary; Measurement: Respondent's answer to the question;
COPD control | 1 year
  Definition: Has the number of acute exacerbations decreased in the past six months?; Variable type: Binary; Measurement: Respondent's answer to the question;
CAT score | 1 year
  Definition: CAT questionnaire for COPD patients; Variable type: Continuous; Measurement: Respondent's answer to the question; Introduction to CAT questionnaire: COPD Assessment Test (CAT) is a questionnaire for people with COPD. It is designed to measure the impact of COPD on a person's life, and how this changes over time. The scope ranges from 0 to 40, the higher the score, the worse the COPD conditions.
mMRC score | 1 year
  Definition: mMRC questionnaire ; Variable type: Categorical; Measurement: Respondent's answer to the question; Introduction to mMRC: Modified Medical Research Council, categorical value, level 0 represents a good respiratory condition, while the maximum level 4 represents a very bad respiratory condition.
Number of outpatient visits | 1 year
  Definition: Outpatient visits and type of hospital; Variable type: Count; Measurement: Insurance/outpatient data/survey data
Number of inpatient visits | 1 year
  Definition: Inpatient visits and type of hospital; Variable type: Count; Measurement: Insurance/inpatient data/survey data
Medical expenditure within a family over the past year | 1 year
  Definition: Healthcare-related expenditures; Variable type: Continuous; Measurement: Survey data/insurance/outpatient/inpatient data;
Depression Symptoms | 1 year
  Definition: Emotional disorders, including sadness, loss, and anger; Variable type: Continuous; Measurement: PHQ-9; Introduction to PHQ-9: Patient Health Questionnaire- 9 items (PHQ-9), ranging from 0 to 27, the higher the score, the severer the depression symptoms for the respondents will be.
Anxiety Symptoms | 1 year
  Definition: Unpleasant state of inner turmoil; Variable type: Continuous; Measurement: GAD-7; Introduction to GAD-7: General Anxiety Disorder - 7 (GAD-7), ranging from 0 to 21, the higher the score, the severer the anxiety symptoms for the respondents will be.
Warwick-Edinburgh Mental Well-being Scale, WEM -WBS score | 1 year
  Definition: Reflects overall mental health problems; Variable type: Continuous; Measurement: WEMWBS; Introduction to WEMWBS: Warwick-Edinburgh Mental Well-being Scale, ranging from 14 to 70, the lower the score, the worse one's general mental health will be.
Blood pressure | 1 year
  Definition: Systolic and diastolic blood pressure (mmHg); Variable type: Continuous; Measurement: Omron portable automatic blood pressure monitor;
Blood Glucose | 1 year
  Definition: Reference standard for average plasma glucose concentration over a period of time; Variable type: Continuous; Measurement: Blood glucose meter;
Waist circumference | 1 year
  Definition: Waist circumference (cm); Variable type: Continuous; Measurement: Soft measuring tape;
BMI | 1 year
  Definition: Body mass index (BMI), weight divided by height squared (kg/m²); Variable type: Continuous; Measurement: Calculation;
Family level annual consumption expenditure | 1 year
  Definition: Annual total household expenditure (self-reported); Variable type: Categorical; Measurement: Answer to a series of questions covering local expenditure categories by the household representative;
Employment status | 1 year
  Definition: Main occupation and type; Variable type: Categorical; Measurement: Respondent's answer to the question;
HBP Screening | 1 year
  Definition: Have you ever had your blood pressure measured by a doctor, nurse, or other healthcare professional?; Variable type: Binary; Measurement: Respondent's answer to the question;
HBP Diagnosis | 1 year
  Definition: Have you ever been diagnosed with hypertension by a doctor?; Variable type: Binary; Measurement: Respondent's answer to the question;
HBP Treatment | 1 year
  Definition: Are you currently taking any antihypertensive medication prescribed by a doctor or other healthcare professional? Variable type: Binary; Measurement: Respondent's answer to the question;
HBP Control | 1 year
  Definition: Blood pressure within the normal range at the end-of-year follow-up; Variable type: Binary; Measurement: Blood pressure measurement;
T2DM Screening | 1 year
  Definition: Have you ever had your blood glucose measured by a doctor, nurse, or other healthcare professional? Variable type: Binary; Measurement: Respondent's answer to the question;
T2DM Diagnosis | 1 year
  Definition: Have you ever been diagnosed with T2DM by a doctor?; Variable type: Binary; Measurement: Respondent's answer to the question;
T2DM Treatment | 1 year
  Definition: Are you currently receiving a type 2 diabetes treatment plan prescribed by a doctor or other healthcare professional?; Variable type: Binary; Measurement: Respondent's answer to the question;
T2DM Control | 1 year
  Definition: Blood glucose within the normal range at the end-of-year follow-up; Variable type: Binary; Measurement: Blood glucose measurement;
Smoking status | 1 year
  Definition: Do you currently smoke? Variable type: Binary/Categorical; Measurement: Respondent's answer to the question;
Smoking Amount | 1 year
  Definition: How many cigarettes do you smoke per day on average?; Variable type: Count; Measurement: Respondent's answer to the question;
Drinking Status | 1 year
  Definition: Frequency of alcohol consumption in the past 3 months; Variable type: Categorical; Measurement: Respondent's answer to the question;
Sugar Consumption | 1 year
  Definition: Frequency of consumption of sugary foods/drinks; Variable type: Categorical; Measurement: Respondent's answer to the question;
Salted Vegetables Consumption | 1 year
  Definition: Frequency of consumption of salty vegetables; Variable type: Categorical; Measurement: Respondent's answer to the question;
Vegetable Consumption | 1 year
  Definition: Frequency of consumption of vegetable; Variable type: Categorical; Measurement: Respondent's answer to the question;
Physical exercise | 1 year
  Definition: Hours of physical exercise per week; Variable type: Count; Measurement: Respondent's answer to the question;
Asthma knowledge | 1 year
  Excerpt of PAKQ, selecting questions that general population should know in terms of asthma, ranging from 0 to 7, the higher the score, the more correct statements the respondents has chosen.
Saint George Respiratory Questionnaire score | 1 year
  Definition: SGRQ questionnaire for COPD patients; Variable type: continuous Measurement: Respondent's answer to the questions; Introduction to SGRQ: Saint George Respiratory Questionnaire score, ranging from 0 to 100, where 0 represents the best possible health status and 100 represents the worst possible health status.
ACT score | 1 year
  Definition: Asthma control test score; Variable type: Continuous; Measurement: Respondent's answer to the questions; Introduction to ACT score: Asthma control test (ACT), ranging from 0 to 25, the lower the score, the better asthma controlled
Asthma diagnosis | 1 year
  Definition: Have you ever diagnosed as asthma patient by professional physician? Variable type: Binary; Measurement: Respondent's answer to the question;
Smoking dependence | 1 year
  Fagerström test for nicotine dependence (FTND) is a scale that measures the nicotine dependence of smokers, ranging from 0 to 15, the higher the value, the worse the nicotine dependence will be. Heaviness Index of Smoking (HIS) could also be calculated using part of the scale, ranging from 0 to 6, and higher score means worse nicotine dependence.
Productivity loss | 1 year
  Working Productivity and Activity Impairment-General Health (WAPI-GH) Chinese version 2.0 is used. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes, as follows:
  Questions:
  1. = currently employed
  2. = hours missed due to health problems
  3. = hours missed other reasons
  4. = hours actually worked
  5. = degree health affected productivity while working
  6. = degree health affected regular activities
  Scores:
  Multiply scores by 100 to express in percentages.
  Percent work time missed due to health: Q2/(Q2+Q4)
  Percent impairment while working due to health: Q5/10
  Percent overall work impairment due to health:
  Q2/(Q2+Q4)+[(1-(Q2/(Q2+Q4)))x(Q5/10)]
  Percent activity impairment due to health: Q6/10

CONTACTS AND LOCATIONS:
Overall Officials: Simiao Chen, Ph.D., Principal Investigator — Peking Union Medical College
Locations (1):
- 26 township hospitals in Xishui County, Zunyi, Guizhou, China

IPD SHARING:
Plan to Share IPD: No